CLINICAL TRIAL: NCT05489263
Title: Derivation and Validation of A Predictive Score System for Acute Kidney Injury Following Pediatric Cardiac Surgery
Brief Title: A Predictive Score System for AKI Following Pediatric Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Jianhui Wang, Department of Anesthesiology, China National Center for Cardiovascular Diseases
Other Study IDs: 2021-LC15
Record Dates: First submitted 2022-03-11; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Congenital Heart Disease; Surgery--Complications; Acute Kidney Injury
Keywords: Pediatric Cardiac Surgery; Acute Kidney Injury; Prediction
MeSH Terms: conditions — Heart Defects, Congenital; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI: AKI is defined by KDIGO criterion based on peri-operative serum creatinine variation.
  Interventions: Other: No intervention
- No-AKI: No-AKI is defined by KDIGO criterion based on peri-operative serum creatinine variation.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Acute kidney injury (AKI) has been recognized as a typical post- operative complication among the children undergoing surgical repair of a congenital cardiac defect. It is associated with increased morbidity and mortality in the intensive care unit and a higher utilization of hospital resources. However, how to precisely identify those who have greater hazard to encounter postoperative AKI seems ambiguous.

DETAILED DESCRIPTION:
The development of AKI is common following cardiac surgery whether in adult or pediatric population. Not only severe AKI like dialysis support, but also mild kidney injury has profound influence on increased subsequent morbidities and mortality.

Pediatric patients who undergo cardiac procedures are characterized by lower weight, younger age, complicated cardiac anomaly and poor resistance to surgical insults. Thus, in comparison with adults, their AKI risk is relatively higher.

At present there has been no specific intervention regarding AKI prevention and therapy. Establishing a risk score based on patient characteristics and surgical information to effectively predict postoperative AKI risk is therefore imperative. It can serve as a decision-making tool to facilitate patient management with regard to kidney prognosis.

This program is aimed at developing and internally validating a AKI risk score post cardiac surgery in a Chinese pediatric population.

ELIGIBILITY:
Inclusion Criteria:

1. < 18 years old
2. Pediatric patients undergoing cardiac surgery in Fuwai Hospital

Exclusion Criteria:

1. Supported by dialysis for renal failure prior to cardiac procedure
2. Previously received a renal transplant
3. Lack of preoperative or postoperative serum creatinine measurements
4. Guardians' refusal on informed consent sign

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A cohort of pediatric patients of 18 years old and younger who have cardiac procedures in Fuwai Hospital, Beijing, China will be consecutively enrolled.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The Prevalence of Acute Kidney Injury | Up to postoperative 7 days
  Acute Kidney Injury was defined by Kidney Disease Improving Global Outcomes (KDIGO) Criteria. Accordingly, AKI was classified as stage 1, stage 2 and stage 3.

SECONDARY OUTCOMES:
The incidence of dialysis | Up to postoperative 7 days
  The therapeutic approach to correct renal failure
The hours of mechanical ventilation | Up to postoperative 7 days
  Time before first extubation
The incidence of reinbutation | Up to hospital discharge, an average of 7 days
  Need for postoperative endotracheal intubation given the occurrence of respiratory or non-respiratory complication after extubation.
The incidence of tracheotomy | Up to hospital discharge, an average of 7 days
  The necessary treatment for postoperative respiratory failure
The incidence of re-operation | Up to hospital discharge, an average of 7 days
  Re-exploration prescribed by surgeons due to cardiac issues or excessive chest drainage volume.
The incidence of mechanical cardiac support | Up to hospital discharge, an average of 7 days
  Supported by extracorporeal membrane oxygenation from operative day to discharge or death
The incidence of mortality | Up to hospital discharge, an average of 7 days
  Specific death reason
The incidence of pulmonary infection | Up to hospital discharge, an average of 7 days
  Assessed by relevant guidelines of pulmonary infection
The cost of medical resources | Up to hospital discharge, an average of 7 days
  The RMB patients spend during the whole hospitalization
Intensive Care Unit Discharge Time | Up to ICU discharge, an average of 5 days
  Time and date when the patient is transferred to ward
Hospital Discharge Time | Up to hospital discharge, an average of 7 days
  Time and date when the patient is discharged from the hospital
The relative change of left ventricular ejection fraction (LVEF) from baseline to hospital discharge | Up to hospital discharge, an average of 7 days
  (LVEF at hospital discharge - LVEF at baseline)/LVEF at baseline * 100%
The relative change of left ventricular end-diastolic diameter (LVEDD) from baseline to hospital discharge | Up to hospital discharge, an average of 7 days
  (LVEDD at hospital discharge - LVEDD at baseline)/LVEDD at baseline * 100%

OTHER OUTCOMES:
The relative change of left ventricular ejection fraction (LVEF) from baseline to postoperative 1 year | Up to postoperative 1 year
  (LVEF at 1 year - LVEF at baseline)/LVEF at baseline * 100%
The relative change of left ventricular end-diastolic diameter (LVEDD) from baseline to postoperative 1 year | Up to postoperative 1 year
  (LVEDD at 1 year - LVEDD at baseline)/LVEDD at baseline * 100%

CONTACTS AND LOCATIONS:
Overall Officials: Jianhui Wang, MD, Principal Investigator — Department of Anesthesiology, Fuwai Hospital, Chinese Academy of Medial Sciences
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
IPD cannot be shared with other researchers. However, data can be provided if requested.

REFERENCES:
- [Derived] Bie D, Li Y, Wang H, Liu Q, Dou D, Jia Y, Yuan S, Li Q, Wang J, Yan F. Relationship between intra-operative urine output and postoperative acute kidney injury in paediatric cardiac surgery: A retrospective observational study. Eur J Anaesthesiol. 2024 Dec 1;41(12):881-888. doi: 10.1097/EJA.0000000000002044. Epub 2024 Aug 16. PMID 39021216